CLINICAL TRIAL: NCT03896295
Title: An Open-label Extension Study of MOM-M281-004 to Evaluate the Safety, Tolerability, and Efficacy of M281 Administered to Patients With Generalized Myasthenia Gravis
Brief Title: An Extension Study of MOM-M281-004 to Evaluate the Safety, Tolerability, and Efficacy of M281 Administered to Patients With Generalized Myasthenia Gravis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was originally halted due to the COVID-19 pandemic. The study was later terminated prematurely as the participants will have the option to enter into an open-label extension portion of a planned future study. It was not due to safety concerns.
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOM-M281-005; 2018-003618-41 (EudraCT Number)
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Generalized Myasthenia Gravis
Keywords: M281; Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M281 (Experimental)
  Interventions: Drug: M281

INTERVENTIONS:
Drug: M281 — M281 injection administered as intravenous infusion

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of M281 in participants with generalized myasthenia gravis (gMG)

ELIGIBILITY:
Participants must be ≥18 years of age with a documented history of Generalized Myasthenia Gravis (gMG) and clinical signs/symptoms of gMG, not pregnant or breastfeeding, previously participated in the MOM-281-004 study, had no major eligibility deviations or other major protocol deviations or not met any of the stopping criteria or discontinued study drug in the MOM-M281-004 study for any reason other than the need for rescue therapy as specified in the MOM-M281-004 study.

Additional, more specific criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (23):
  - Momenta Investigational Site, Phoenix, Arizona
  - Momenta Investigational Site, Los Angeles, California
  - Momenta Investigational Site, Orange, California
  - Momenta Investigational Site, Stanford, California
  - Momenta Investigational Site, Aurora, Colorado
  - Momenta Investigational Site, New Haven, Connecticut
  - Momenta Investigational Site, Boca Raton, Florida
  - Momenta Investigational Site, Maitland, Florida
  - Momenta Investigational Site, Port Charlotte, Florida
  - Momenta Investigational Site, St. Petersburg, Florida
  - Momenta Investigational Site, Augusta, Georgia
  - Momenta Investigational Site, Fairway, Kansas
  - Momenta Investigational Site, Boston, Massachusetts
  - Momenta Investigational Site, New Brunswick, New Jersey
  - Momenta Investigational Site, New York, New York
  - Momenta Investigational Site, Charlotte, North Carolina
  - Momenta Investigational Site, Durham, North Carolina
  - Momenta Investigational Site, Raleigh, North Carolina
  - Momenta Investigational Site, Cincinnati, Ohio
  - Momenta Investigational Site, Columbus, Ohio
  - Momenta Investigational Site, Cordova, Tennessee
  - Momenta Investigational Site, Austin, Texas
  - Momenta Investigational Site, Round Rock, Texas
- Belgium (3):
  - Momenta Investigational Site, Leuven, Vlaams Brabant
  - Momenta Investigational Site, Antwerp
  - Momenta Investigational Site, Brussels
- Canada (4):
  - Momenta Investigational Site, Edmonton, Alberta
  - Momenta Investigational Site, London, Ontario
  - Momenta Investigational Site, Toronto, Ontario
  - Momenta Investigational Site, Québec, Quebec
- Germany (4):
  - Momenta Investigational Site, Göttingen, Lower Saxony
  - Momenta Investigational Site, Düsseldorf
  - Momenta Investigational Site, Gummersbach
  - Momenta Investigational Site, Münster
- Italy (3):
  - Momenta Investigational Site, Cefalù
  - Momenta Investigational Site, Messina
  - Momenta Investigational Site, Milan
- Poland (3):
  - Momenta Investigational Site, Krakow
  - Momenta Investigational Site, Lodz
  - Momenta Investigational Site, Warsaw
- Spain (7):
  - Momenta Investigational Site, Barcelona, Catalan
  - Momenta Investigational Site, Barcelona, Catalonia
  - Momenta Investigational Site, L'Hospitalet de Llobregat, Catalonia
  - Momenta Investigational Site, Donostia / San Sebastian, Gipuzkoa
  - Momenta Investigational Site, Madrid
  - Momenta Investigational Site, Seville
  - Momenta Investigational Site, Valencia
- United Kingdom (2):
  - Momenta Investigational Site, Birmingham
  - Momenta Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from study MOM-M281-004 (NCT03772587) who completed the Day 113 visit of that study were eligible to enroll in this open-label extension study (MOM-M281-005). The Day 113 visit of MOM-M281-004 occurred approximately 8 weeks after the last dose in that study.
Groups:
- Placebo-Nipocalimab: Participants who received placebo in MOM-M281-004 (NCT03772587) study rolled-over and received intravenous (IV) infusion of nipocalimab (M281) 30 milligrams per kilogram (mg/kg) every 4 weeks (Q4W) starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding every 2 weeks (Q2W).
- Nipocalimab-Nipocalimab: Participants who received nipocalimab in MOM-M281-004 study rolled-over and received IV infusion of nipocalimab 30 mg/kg Q4W starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding Q2W.
Period: Overall Study
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab
Started | 7 | 30
Completed | 0 | 0
Not Completed | 7 | 30
Not completed — Adverse Event | 0 | 1
Not completed — COVID-19 | 7 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Total
Number analyzed (Participants) | 7 | 30 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 20 | 25
  >=65 years | 2 | 10 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (20.39) | 53 (16.93) | 53.2 (17.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 18 | 22
  Male | 3 | 12 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 28 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 5 | 29 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  GERMANY | 1 | 1 | 2
  ITALY | 0 | 2 | 2
  POLAND | 0 | 7 | 7
  SPAIN | 4 | 7 | 11
  UNITED STATES | 2 | 13 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as any AE occurring during or after the initiation of the first infusion of study drug in this study.
Time Frame: Up to 257 days post-baseline (Baseline is Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo-Nipocalimab: Participants who received placebo in MOM-M281-004 study rolled-over and received intravenous (IV) infusion of nipocalimab 30 milligrams per kilogram (mg/kg) every 4 weeks (Q4W) starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding every 2 weeks (Q2W).
- Nipocalimab (All Participants): Participants who received placebo or nipocalimab in MOM-M281-004 study rolled-over and received IV infusion of nipocalimab 30 mg/kg Q4W starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding Q2W.
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 30 | 37
Participants | 4 | 18 | 22

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. SAE is defined as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
Time Frame: Up to 257 days post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Placebo-Nipocalimab: Participants who received placebo in MOM-M281-004 study rolled-over and received IV infusion of nipocalimab 30 mg/kg every Q4W starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding Q2W.
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 30 | 37
Participants | 1 | 4 | 5

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (AESIs)
Description: Number of participants with treatment-emergent AESIs were reported. Severe infections and hypoalbuminemia (Grade 3 or higher according to the Common Terminology Criteria for Adverse Events [CTCAE] v5.0) were considered as AESIs.
Time Frame: Up to 257 days post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Nipocalimab (All Participants): All participants who received placebo or nipocalimab in MOM-M281-004 study rolled-over and received IV infusion of nipocalimab 30 mg/kg Q4W starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding Q2W.
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 30 | 37
Participants | 1 | 1 | 2

4. Primary Outcome: Number of Participants With Treatment-emergent Abnormal Vital Signs
Description: Number of participants with treatment-emergent abnormal vital signs including pulse rate (less than or equal to [<=] 50 beats per minutes [bpm] with greater than or equal to [>=] 15 bpm decrease from baseline, >= 120 bpm with >=15 bpm increase from baseline), systolic blood pressure (SBP) (<= 90 millimeters of mercury [mmHg] with >= 20 mmHg decrease from baseline, >= 160 mmHg with >= 20 mmHg increase from baseline) and diastolic blood pressure (DBP) (<= 50 mmHg with >=15 mmHg decrease from baseline, >=100 mmHg with >=15 mmHg decrease from baseline) were reported.
Time Frame: Up to 257 days post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 30 | 37
Participants
  Pulse rate: <=50 bpm with >=15 bpm decrease from baseline | 0 | 0 | 0
  Pulse rate: >= 120 bpm with >=15 bpm increase from baseline | 0 | 0 | 0
  SBP: <= 90 mmHg with >= 20 mmHg decrease from baseline | 0 | 1 | 1
  SBP: >= 160 mmHg with >= 20 mmHg increase from baseline | 0 | 1 | 1
  DBP: <= 50 mmHg with >=15 mmHg decrease from baseline | 0 | 2 | 2
  DBP: >=100 mmHg with >=15 mmHg decrease from baseline | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormalities in Physical Examinations
Description: Number of participants with abnormalities in physical examinations (abdomen, head, ears, eyes, nose, throat, and sinuses, lungs, neurological, skin, blood and lymphatic system, cardiovascular, chest, gastrointestinal, general appearance and musculoskeletal) were reported.
Time Frame: Week 12
Population: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this outcome measure (OM). Here, 'n' (number analyzed) specifies the number of participants evaluated for specific categories. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
Participants
  Abdomen | 1 | 0 | 1
  Head, Ears, Eyes, Nose, Throat and Sinuses | 0 | 0 | 0
  Lungs | 0 | 0 | 0
  Neurological: number analyzed (Participants) | 4 | 16 | 20
  Neurological | 0 | 1 | 1
  Skin | 1 | 4 | 5

6. Primary Outcome: Change From Baseline in Chemistry Laboratory Parameters: Albumin and Protein
Description: Change from baseline in chemistry laboratory parameters: albumin and protein were reported.
Time Frame: Baseline up to Week 12
Population: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this outcome measure (OM). As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Groups:
- Placebo-Nipocalimab: Participants who received placebo in MOM-M281-004 study rolled-over and received IV infusion of nipocalimab 30 mg/kg Q4W starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding Q2W.
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
grams per liter (g/L)
  Albumin | -1.5 (2.89) | -1.2 (3.21) | -1.3 (3.08)
  Protein | -3.5 (2.08) | -3.8 (4.99) | -3.7 (4.54)

7. Primary Outcome: Change From Baseline in Chemistry Laboratory Parameters: Bicarbonate, Calcium, Chloride, Cholesterol, Glucose, Phosphate, Potassium, Sodium, Triglycerides, Urate and Urea Nitrogen
Description: Change from baseline in chemistry laboratory parameters: bicarbonate, calcium, chloride, cholesterol, glucose, phosphate, potassium, sodium, triglycerides, urate and urea nitrogen were reported.
Time Frame: Baseline up to Week 12
Population: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
millimoles per liter (mmol/L)
  Bicarbonate | -2.0 (2.45) | 1.6 (2.91) | 1.0 (3.14)
  Calcium | 0.010 (0.0627) | -0.018 (0.1005) | -0.013 (0.0938)
  Chloride | 0.5 (1.91) | 0.6 (2.85) | 0.6 (2.66)
  Cholesterol | 0.480 (1.0100) | 0.261 (0.5732) | 0.303 (0.6509)
  Glucose | 0.280 (0.5054) | -0.258 (1.1401) | -0.155 (1.0607)
  Phosphate | -0.018 (0.0971) | -0.002 (0.1903) | -0.005 (0.1744)
  Potassium | 0.05 (0.173) | 0.05 (0.583) | 0.05 (0.526)
  Sodium | 0.8 (0.96) | 1.4 (2.18) | 1.2 (2.00)
  Triglycerides | 0.223 (0.5799) | 0.081 (0.3223) | 0.108 (0.3699)
  Urate | -0.0090 (0.04285) | 0.0174 (0.04790) | 0.124 (0.04716)
  Urea Nitrogen | -0.270 (1.7830) | -0.105 (1.7292) | -0.136 (1.6951)

8. Primary Outcome: Change From Baseline in Chemistry Laboratory Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Creatine Kinase, Gamma Glutamyl Transferase, Lactate Dehydrogenase
Description: Change from baseline in chemistry laboratory parameters alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), creatine kinase, gamma glutamyl transferase, lactate dehydrogenase were reported.
Time Frame: Baseline up to Week 12
Population: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific categories. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
units per liter (U/L)
  ALT | 17.0 (28.76) | 2.6 (5.33) | 5.3 (13.43)
  Alkaline Phosphatase: number analyzed (Participants) | 4 | 16 | 20
  Alkaline Phosphatase | 6.3 (2.06) | 5.2 (11.46) | 5.4 (10.23)
  AST | 23.5 (47.67) | 0.9 (3.42) | 5.2 (20.80)
  Creatine Kinase | -17.8 (33.13) | 13.6 (38.34) | 7.7 (38.73)
  Gamma Glutamyl Transferase | 4.3 (11.95) | 1.5 (13.21) | 2.0 (12.74)
  Lactate Dehydrogenase: number analyzed (Participants) | 4 | 16 | 20
  Lactate Dehydrogenase | 30.0 (15.68) | 30.9 (58.10) | 30.7 (52.00)

9. Primary Outcome: Change From Baseline in Chemistry Laboratory Parameters: Bilirubin, Creatinine and Direct Bilirubin
Description: Change from baseline in chemistry laboratory parameters: bilirubin, creatinine and direct bilirubin were reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micromoles per liter (micromol/L)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
micromoles per liter (micromol/L)
  Bilirubin | 0.13 (2.616) | -0.59 (2.403) | -0.46 (2.393)
  Creatinine | -9.0 (7.35) | -2.6 (13.20) | -3.9 (12.41)
  Direct Bilirubin: number analyzed (Participants) | 1 | 2 | 3
  Direct Bilirubin | -1.20 (NA) — Here, NA indicates that standard deviation cannot be calculated for 1 participant. | -0.70 (0.283) | -0.87 (0.359)

10. Primary Outcome: Change From Baseline in Hematology Laboratory Parameter: Erythrocytes (Red Blood Cell)
Description: Change from baseline in erythrocytes (red blood cells) (hematology laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^12 cells count per Liter
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
10^12 cells count per Liter | 0.188 (0.0822) | 0.121 (0.2702) | 0.135 (0.2438)

11. Primary Outcome: Change From Baseline in Hematology Laboratory Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Change from baseline in hematology laboratory parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes were reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells count per Liter
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
10^9 cells count per Liter
  Basophils: number analyzed (Participants) | 4 | 8 | 12
  Basophils | -0.003 (0.0150) | 0.010 (0.0200) | 0.006 (0.0188)
  Eosinophils: number analyzed (Participants) | 4 | 13 | 17
  Eosinophils | 0.015 (0.0465) | 0.013 (0.0776) | 0.014 (0.0702)
  Lymphocytes | -0.045 (0.4498) | 0.063 (0.4715) | 0.041 (0.4576)
  Monocytes | -0.105 (0.1964) | 0.059 (0.2008) | 0.027 (0.2061)
  Neutrophils | -0.433 (0.5744) | 0.411 (1.8622) | 0.243 (1.7058)
  Platelets | 27.8 (11.81) | 12.3 (53.20) | 15.4 (47.93)
  Leukocytes | -0.568 (0.9214) | 0.567 (1.9956) | 0.340 (1.8694)

12. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration
Description: Change from baseline in erythrocytes mean corpuscular hemoglobin (HGB) concentration (hematology laboratory parameter) were reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
grams per Liter (g/L) | -6.5 (25.70) | -2.1 (7.61) | -3.0 (12.38)

13. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin (HGB)
Description: Change from baseline in erythrocytes mean corpuscular HGB (hematology laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
picograms (pg) | 0.03 (0.873) | -0.61 (0.813) | -0.48 (0.842)

14. Primary Outcome: Change From Baseline in Hematology Laboratory Parameter: Erythrocytes Mean Corpuscular Volume
Description: Change from baseline in erythrocytes mean corpuscular volume (hematology laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
femtoliters (fL) | 2.45 (6.174) | -1.41 (3.406) | -0.64 (4.206)

15. Primary Outcome: Change From Baseline in Hematology Laboratory Parameter: Hematocrit
Description: Change from baseline in hematocrit (hematology laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liter of cells per liter of blood (L/L)
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
liter of cells per liter of blood (L/L) | 0.0278 (0.03542) | 0.0048 (0.02401) | 0.0094 (0.02725)

16. Primary Outcome: Change From Baseline in Hematology Laboratory Parameter: Hemoglobin
Description: Change from baseline in hemoglobin (hematology laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 16 | 20
g/L | 5.8 (4.65) | 0.6 (7.29) | 1.7 (7.06)

17. Primary Outcome: Change From Baseline in Urinalysis Laboratory Parameter: pH
Description: Change from baseline in pH (urinalysis laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
pH | -0.8 (0.96) | 0.0 (1.06) | -0.1 (1.06)

18. Primary Outcome: Change From Baseline in Urinalysis Laboratory Parameter: Specific Gravity
Description: Change from baseline in specific gravity (urinalysis laboratory parameter) was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 17 | 21
ratio | -0.0003 (0.00660) | -0.0030 (0.00973) | -0.0025 (0.00914)

19. Primary Outcome: Number of Participants With Treatment-emergent Abnormal Electrocardiograms (ECG) Values
Description: Number of participants with treatment-emergent abnormal ECG values for variables including mean heart rate (abnormally low refers to less than or equal to [<=] 50 beats per minute [bpm], abnormally high refers greater than or equal to [>=] 120 bpm), PR interval (abnormally low refers to < 120 and abnormally high refers to >200 milliseconds [msec]), RR interval (abnormally low refers to <600 msec and abnormally high refers to >1200 msec) and QRS duration (abnormally > 120) were reported.
Time Frame: Up to 257 days post-baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Placebo-Nipocalimab: Participants who received placebo in MOM-M281-004 study rolled-over and received IV infusion of nipocalimab 30 mg/kg every Q4W starting Day 1 up to 8 weeks. After 8 weeks of treatment on a stable dose of nipocalimab, the dose and/or dosing frequency could be individually adjusted, at the investigator's discretion to receive maximum dose of 60 mg/kg at a frequency of not exceeding every Q2W.
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 29 | 36
Participants
  ECG Mean Heart Rate (<= 50) | 0 | 5 | 5
  ECG Mean Heart Rate (>=120) | 0 | 0 | 0
  PR Interval (<120) | 0 | 0 | 0
  PR Interval (> 200) | 0 | 5 | 5
  RR Interval (<600) | 0 | 0 | 0
  RR Interval (>=1200) | 0 | 4 | 4
  QRS Duration (>120) | 1 | 3 | 4

20. Primary Outcome: Number of Participants With Columbia Suicide Severity Rating Scale (C-SSRS) Scores
Description: Number of participants with C-SSRS scores were reported. C-SSRS is a clinician-administered questionnaire designed to solicit occurrence, severity, and frequency of suicide-related ideation and behaviors. Total score ranges from 1 to 10, score of 0 was assigned (0="no event that can be assessed based on C-SSRS"). Higher total scores indicate greater severity. Maximum score assigned for each participant was summarized into one of 3 categories: no suicidal ideation or behavior (0), suicidal ideation (1 to 5): higher score indicates more suicidal ideation, suicidal behavior (6 to 10): higher score indicates more suicidal behavior. Suicidal ideation includes participants who did not have suicidal ideation or behavior at baseline and had suicidal ideation without behavior at some time point post-baseline. Suicidal behavior includes participants who did not have suicidal ideation or behavior at baseline and had suicidal behavior at some time point post-baseline (baseline=Day 1).
Time Frame: Up to 257 days post-baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 6 | 30 | 36
Participants
  No Suicidal Ideation/Behavior | 5 | 30 | 35
  Suicidal Ideation | 1 | 0 | 1
  Suicidal Behavior | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in Total Myasthenia Gravis - Activities of Daily Living (MG-ADL) Score Over Time
Description: The MG-ADL was used to assess the participant's MG symptom severity. It assesses eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, and eyelid droop) which were rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score is the sum of the eight function scores and ranges from 0 to 24. Higher scores indicated greater symptom severity/difficulty in performing daily living activities.
Time Frame: Baseline up to Weeks 4, 8, 12, 24, End of treatment (EoT) (up to 253 days post-baseline), Follow-up (up to 257 days post-baseline)
Population: The full analysis set (FAS) included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific timepoints. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 5 | 26 | 31
score on a scale
  Week 4 | 0.6 (1.34) | -0.6 (2.42) | -0.4 (2.30)
  Week 8: number analyzed (Participants) | 5 | 19 | 24
  Week 8 | -0.8 (3.70) | -0.9 (2.63) | -0.9 (2.80)
  Week 12: number analyzed (Participants) | 4 | 17 | 21
  Week 12 | -0.3 (4.35) | -1.2 (2.49) | -1.0 (2.82)
  Week 24: number analyzed (Participants) | 1 | 5 | 6
  Week 24 | -1.0 (NA) — Here, NA indicates that standard deviation could not be calculated for 1 participant. | -1.2 (1.92) | -1.2 (1.72)
  EoT (up to 253 days post-baseline): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline) |  | -2.4 (2.55) | -2.4 (2.55)
  Follow-up (up to 257 days post-baseline): number analyzed (Participants) | 5 | 24 | 29
  Follow-up (up to 257 days post-baseline) | -0.6 (1.14) | 1.2 (3.08) | 0.9 (2.91)

22. Secondary Outcome: Number of Participants With a 2-, 3-, 4-, 5-, 6-, 7-, or Greater Than or Equal to (>=) 8-point Improvement in Total MG-ADL Score Over Time
Description: Number of Participants With a 2-, 3-, 4-, 5-, 6-, 7-, or greater than or equal to (>=) 8-point improvement in total MG-ADL score over time were reported. MG-ADL was used to assess the participant's MG symptom severity. It assesses eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, and eyelid droop) which were rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score is the sum of the eight function scores and ranges from 0 to 24. Higher scores indicated greater symptom severity/difficulty in performing daily living activities.
Time Frame: Weeks 4, 8, 12, 24, End of treatment (EoT) (up to 253 days post-baseline), Follow-up (up to 257 days post-baseline)
Population: The FAS included all participants who received at least 1 dose of study drug nipocalimab. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific timepoints. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 30 | 37
Participants
  Week 4 (2 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (2 Point Improvement) |  | 2 | 2
  Week 4 (3 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (3 Point Improvement) |  | 1 | 1
  Week 4 (4 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (4 Point Improvement) |  | 0 | 0
  Week 4 (5 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (5 Point Improvement) |  | 1 | 1
  Week 4 (6 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (6 Point Improvement) |  | 2 | 2
  Week 4 (7 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (7 Point Improvement) |  | 0 | 0
  Week 4 (>= 8 Point Improvement): number analyzed (Participants) | 0 | 6 | 6
  Week 4 (>= 8 Point Improvement) |  | 0 | 0
  Week 8 (2 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (2 Point Improvement) | 1 | 2 | 3
  Week 8 (3 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (3 Point Improvement) | 0 | 4 | 4
  Week 8 (4 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (4 Point Improvement) | 0 | 0 | 0
  Week 8 (5 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (5 Point Improvement) | 0 | 0 | 0
  Week 8 (6 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (6 Point Improvement) | 1 | 0 | 1
  Week 8 (7 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (7 Point Improvement) | 0 | 0 | 0
  Week 8 (>= 8 Point Improvement): number analyzed (Participants) | 2 | 7 | 9
  Week 8 (>= 8 Point Improvement) | 0 | 1 | 1
  Week 12 (2 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (2 Point Improvement) | 0 | 2 | 2
  Week 12 (3 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (3 Point Improvement) | 0 | 0 | 0
  Week 12 (4 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (4 Point Improvement) | 0 | 0 | 0
  Week 12 (5 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (5 Point Improvement) | 0 | 0 | 0
  Week 12 (6 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (6 Point Improvement) | 1 | 3 | 4
  Week 12 (7 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (7 Point Improvement) | 0 | 0 | 0
  Week 12 (>= 8 Point Improvement): number analyzed (Participants) | 1 | 5 | 6
  Week 12 (>= 8 Point Improvement) | 0 | 0 | 0
  Week 24 (2 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (2 Point Improvement) |  | 1 | 1
  Week 24 (3 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (3 Point Improvement) |  | 0 | 0
  Week 24 (4 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (4 Point Improvement) |  | 1 | 1
  Week 24 (5 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (5 Point Improvement) |  | 0 | 0
  Week 24 (6 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (6 Point Improvement) |  | 0 | 0
  Week 24 (7 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (7 Point Improvement) |  | 0 | 0
  Week 24 (>= 8 Point Improvement): number analyzed (Participants) | 0 | 2 | 2
  Week 24 (>= 8 Point Improvement) |  | 0 | 0
  EoT (up to 253 days post-baseline) (2 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (2 Point Improvement) |  | 2 | 2
  EoT (up to 253 days post-baseline) (3 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (3 Point Improvement) |  | 2 | 2
  EoT (up to 253 days post-baseline) (4 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (4 Point Improvement) |  | 0 | 0
  EoT (up to 253 days post-baseline) (5 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (5 Point Improvement) |  | 1 | 1
  EoT (up to 253 days post-baseline) (6 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (6 Point Improvement) |  | 1 | 1
  EoT (up to 253 days post-baseline) (7 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (7 Point Improvement) |  | 2 | 2
  EoT (up to 253 days post-baseline) (>= 8 Point Improvement): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline) (>= 8 Point Improvement) |  | 0 | 0
  Follow-up (up to 257 days post-baseline) (2 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (2 Point Improvement) | 1 | 3 | 4
  Follow-up (up to 257 days post-baseline) (3 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (3 Point Improvement) | 0 | 1 | 1
  Follow-up (up to 257 days post-baseline) (4 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (4 Point Improvement) | 0 | 0 | 0
  Follow-up (up to 257 days post-baseline) (5 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (5 Point Improvement) | 0 | 0 | 0
  Follow-up (up to 257 days post-baseline) (6 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (6 Point Improvement) | 0 | 0 | 0
  Follow-up (up to 257 days post-baseline) (7 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (7 Point Improvement) | 0 | 0 | 0
  Follow-up (up to 257 days post-baseline) (>= 8 Point Improvement): number analyzed (Participants) | 1 | 4 | 5
  Follow-up (up to 257 days post-baseline) (>= 8 Point Improvement) | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Total Quantitative Myasthenia Gravis (QMG) Score Over Time
Description: The QMG test was used to assess the participant's strength. The quantitative results of each of the 13 strength components were mapped to a 4-point scale where 0 equals to (=) none, 1= mild, 2= moderate and 3= severe. The total score is the sum of the 13 scale scores and ranges from 0 to 39. Higher scores indicated more severe impairment.
Time Frame: as for outcome 21
Population: The FAS included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific timepoints. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 2 | 9 | 11
score on a scale
  Week 4 | 1.5 (6.36) | -1.3 (2.60) | -0.8 (3.28)
  Week 8: number analyzed (Participants) | 2 | 7 | 9
  Week 8 | -3.0 (5.66) | 1.0 (1.53) | 0.1 (2.98)
  Week 12: number analyzed (Participants) | 2 | 6 | 8
  Week 12 | -0.5 (3.54) | -1.2 (2.23) | -1.0 (2.33)
  Week 24: number analyzed (Participants) | 0 | 3 | 3
  Week 24 |  | -2.7 (1.53) | -2.7 (1.53)
  EoT (up to 253 days post-baseline): number analyzed (Participants) | 0 | 7 | 7
  EoT (up to 253 days post-baseline) |  | -2.4 (4.12) | -2.4 (4.12)
  Follow-up (up to 257 days post-baseline): number analyzed (Participants) | 1 | 7 | 8
  Follow-up (up to 257 days post-baseline) | -3.0 (NA) — Here, NA indicates that standard deviation could not be calculated for 1 participant. | -1.6 (2.07) | -1.8 (1.98)

24. Secondary Outcome: Change From Baseline in Total Revised Myasthenia Gravis Quality of Life - 15 Scale (MG-QoL15r) Score Over Time
Description: The MG-QoL15r was used to assess the participant's limitations related to living with MG. It consists of 15 questions and each of the 15 questions were rated by the participant on a 3-point scale (0= Not at all, 1= somewhat, 2=very much) based on a recall period of "over the past few weeks". The total score is the sum of the 15 question scores and ranges from 0 to 30. Higher scores indicated more limitation.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 30 | 37
score on a scale
  Week 4: number analyzed (Participants) | 5 | 26 | 31
  Week 4 | 1.4 (3.85) | -2.2 (4.53) | -1.6 (4.57)
  Week 8: number analyzed (Participants) | 5 | 19 | 24
  Week 8 | -0.4 (3.97) | -1.9 (4.34) | -1.6 (4.23)
  Week 12: number analyzed (Participants) | 4 | 17 | 21
  Week 12 | -1.0 (6.27) | -3.4 (4.70) | -2.9 (4.95)
  Week 24: number analyzed (Participants) | 1 | 5 | 6
  Week 24 | -3.0 (NA) — Here, NA indicates that standard deviation could not be calculated for 1 participant. | -1.4 (1.52) | -1.7 (1.51)
  EoT (up to 253 days post-baseline): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline) |  | -3.7 (5.28) | -3.7 (5.28)
  Follow-up (up to 257 days post-baseline): number analyzed (Participants) | 6 | 24 | 30
  Follow-up (up to 257 days post-baseline) | -1.3 (5.72) | 0.1 (3.11) | -0.2 (3.69)

25. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Rating Score Over Time
Description: The CGI-S scale is the clinician/physician's global assessment of participants illness severity of MG and is rated by answering on 8-point scale. Considering total clinical experience, participant is assessed on severity of illness according to: 0=not performed; 1=normal, not at all ill; 2=borderline illness; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill patients. Higher scores indicated more severity of illness. Values of 0 (not assessed) were excluded from analysis. CGI-S permits global evaluation of participant's condition at given time.
Time Frame: as for outcome 21
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 5 | 26 | 31
score on a scale
  Week 4 | -0.2 (0.84) | -0.3 (0.60) | -0.3 (0.63)
  Week 8: number analyzed (Participants) | 5 | 19 | 24
  Week 8 | -1.0 (0.71) | -0.6 (0.90) | -0.7 (0.86)
  Week 12: number analyzed (Participants) | 4 | 17 | 21
  Week 12 | -0.5 (1.00) | -0.5 (0.80) | -0.5 (0.81)
  Week 24: number analyzed (Participants) | 1 | 5 | 6
  Week 24 | 0.0 (NA) — Here, NA indicates that standard deviation could not be calculated for 1 participant. | -0.6 (0.89) | -0.5 (0.84)
  EoT (up to 253 days post-baseline): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline) |  | -0.7 (0.95) | -0.7 (0.95)
  Follow-up (up to 257 days post-baseline): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) | -1.0 (1.22) | -0.1 (0.73) | -0.3 (0.88)

26. Secondary Outcome: Number of Participants With Improvement of Illness Over Time Based on Clinical Global Impression of Improvement (CGI-I) Scale Score
Description: Number of participants with improvement of illness based on CGI-I scale score over time were reported. The CGI-I scale is the clinician/physician's global assessment of the change in severity of the patient's generalized myasthenia gravis (gMG) since starting this study. The rating is given on a 7-point scale with lower scores indicating greater improvement (1= Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 =Minimally worse; 6 = Much worse; 7 = Very much worse. Values of 0 (not assessed) were excluded from analysis. Higher score indicates more severity.
Time Frame: Weeks 4, 8, 12, 24, End of Treatment (EoT) (up to 253 days post-baseline), Follow-up (up to 257 days post-baseline)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 5 | 26 | 31
Participants
  Week 4 (Very much worse) | 0 | 0 | 0
  Week 4 (Much worse) | 0 | 0 | 0
  Week 4 (Minimally worse) | 1 | 2 | 3
  Week 4 (No change) | 1 | 7 | 8
  Week 4 (Minimally improved) | 2 | 12 | 14
  Week 4 (Much improved) | 0 | 5 | 5
  Week 4 (Very much improved) | 1 | 0 | 1
  Week 8 (Very much worse): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (Very much worse) | 0 | 0 | 0
  Week 8 (Much worse): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (Much worse) | 0 | 0 | 0
  Week 8 (Minimally worse): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (Minimally worse) | 0 | 2 | 2
  Week 8 (No change): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (No change) | 0 | 3 | 3
  Week 8 (Minimally improved): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (Minimally improved) | 2 | 6 | 8
  Week 8 (Much improved): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (Much improved) | 2 | 8 | 10
  Week 8 (Very much improved): number analyzed (Participants) | 5 | 19 | 24
  Week 8 (Very much improved) | 1 | 0 | 1
  Week 12 (Very much worse): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (Very much worse) | 0 | 0 | 0
  Week 12 (Much worse): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (Much worse) | 0 | 0 | 0
  Week 12 (Minimally worse): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (Minimally worse) | 0 | 2 | 2
  Week 12 (No change): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (No change) | 2 | 1 | 3
  Week 12 (Minimally improved): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (Minimally improved) | 1 | 3 | 4
  Week 12 (Much improved): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (Much improved) | 1 | 10 | 11
  Week 12 (Very much improved): number analyzed (Participants) | 4 | 17 | 21
  Week 12 (Very much improved) | 0 | 1 | 1
  Week 24 (Very Much worse): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (Very Much worse) | 0 | 0 | 0
  Week 24 (Much worse): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (Much worse) | 0 | 0 | 0
  Week 24 (Minimally worse): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (Minimally worse) | 0 | 0 | 0
  Week 24 (No change): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (No change) | 1 | 0 | 1
  Week 24 (Minimally improved): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (Minimally improved) | 0 | 1 | 1
  Week 24 (Much improved): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (Much improved) | 0 | 4 | 4
  Week 24 (Very Much improved): number analyzed (Participants) | 1 | 5 | 6
  Week 24 (Very Much improved) | 0 | 0 | 0
  EoT (up to 253 days post-baseline)(Very Much worse): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline)(Very Much worse) |  | 0 | 0
  EoT (up to 253 days post-baseline)(Much worse): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline)(Much worse) |  | 0 | 0
  EoT (up to 253 days post-baseline) (Minimally worse): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline) (Minimally worse) |  | 0 | 0
  EoT (up to 253 days post-baseline) (No change): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline) (No change) |  | 1 | 1
  EoT (up to 253 days post-baseline)(Minimally improved): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline)(Minimally improved) |  | 7 | 7
  EoT (up to 253 days post-baseline)(Much improved): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline)(Much improved) |  | 7 | 7
  EoT (up to 253 days post-baseline)(Very much improved): number analyzed (Participants) | 0 | 16 | 16
  EoT (up to 253 days post-baseline)(Very much improved) |  | 1 | 1
  Follow-up (up to 257 days post-baseline) (Very Much worse): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (Very Much worse) | 0 | 0 | 0
  Follow-up (up to 257 days post-baseline) (Much worse): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (Much worse) | 1 | 2 | 3
  Follow-up (up to 257 days post-baseline) (Minimally worse): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (Minimally worse) | 0 | 3 | 3
  Follow-up (up to 257 days post-baseline) (No change): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (No change) | 0 | 5 | 5
  Follow-up (up to 257 days post-baseline) (Minimally improved): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (Minimally improved) | 0 | 8 | 8
  Follow-up (up to 257 days post-baseline) (Much improved): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (Much improved) | 3 | 2 | 5
  Follow-up (up to 257 days post-baseline) (Very much improved): number analyzed (Participants) | 5 | 21 | 26
  Follow-up (up to 257 days post-baseline) (Very much improved) | 1 | 1 | 2

27. Secondary Outcome: Number of Participants With Change From Baseline in Myasthenia Gravis Foundation of America (MGFA) Classification Score Over Time
Description: Number of participants with change from baseline in MGFA classification score over time were reported. The MGFA was used to assess the participant's MG severity. MGFA classification identifies the subgroup participants with MG who share distinct clinical features or severity of disease: Class I (ocular MG), classes II, III and IV generalized MG with mild, moderate and severe disease, respectively; Class V MG crisis. Separate subclasses under classes II, III and IV are designed: "a" if the predominant weakness is affecting limb/axial weakness or both; subclass "b" if the predominant weakness is affecting oropharyngeal or respiratory muscles or both. In the MGFA classification, lower roman numerals mean less severity. Changes in MGFA classification (regardless of subclass) are categorized as "Improved" (example, III to II), "Same" (example, II to II), or "Worsened" (example, II to III).
Time Frame: Weeks 8, 24 and End of Treatment (EoT) (up to 253 days post-baseline)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 4 | 9 | 13
Participants
  Week 8 (Improved) | 1 | 5 | 6
  Week 8 (Same) | 3 | 3 | 6
  Week 8 (Worsened) | 0 | 1 | 1
  Week 24 (Improved): number analyzed (Participants) | 1 | 1 | 2
  Week 24 (Improved) | 0 | 0 | 0
  Week 24 (Same): number analyzed (Participants) | 1 | 1 | 2
  Week 24 (Same) | 1 | 1 | 2
  Week 24 (Worsened): number analyzed (Participants) | 1 | 1 | 2
  Week 24 (Worsened) | 0 | 0 | 0
  EoT (up to 253 days post-baseline)(Improved): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline)(Improved) |  | 4 | 4
  EoT (up to 253 days post-baseline)(Same): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline)(Same) |  | 3 | 3
  EoT (up to 253 days post-baseline)(Worsened): number analyzed (Participants) | 0 | 8 | 8
  EoT (up to 253 days post-baseline)(Worsened) |  | 1 | 1

28. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to Nipocalimab
Description: Number of participants with ADA to nipocalimab were reported. The presence of ADA to nipocalimab in serum was determined by a sensitive and drug-tolerant electrochemiluminescence immunoassay (ECLIA) method.
Time Frame: Up to 257 days post-baseline
Population: The FAS included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 6 | 29 | 35
Participants | 1 | 16 | 17

29. Secondary Outcome: Number of Participants With Neutralizing Antibodies (NAbs) to Nipocalimab
Description: Number of participants with NAbs were reported. Neutralizing antibodies to nipocalimab were assessed using a non-cell based competitive ligand binding ECLIA assay.
Time Frame: Up to 257 days post-baseline
Population: FAS included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were positive for antibodies to nipocalimab. Per planned analysis, both individual arms and an arm for all (total) participants is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 1 | 16 | 17
Participants | 0 | 4 | 4

30. Primary Outcome: Number of Participants With Below/Above Normal Values of Coagulation Laboratory Parameter
Description: Number of participants with at least one value above upper limit of normal (>ULN) or below the lower limit of normal (< LLN) value of coagulation parameters (activated partial thromboplastin time [APTT] and prothrombin time [PT]) were reported. The lab reference range for APTT is 25.1 to 36.5 seconds. The lab reference range for PT is 9.4 to 12.5 seconds.
Time Frame: Up to 257 days post-baseline
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 7 | 28 | 35
Participants
  APTT (>ULN) | 2 | 15 | 17
  APTT (<LLN) | 0 | 3 | 3
  PT (>ULN) | 1 | 8 | 9
  PT (<ULN) | 0 | 1 | 1

31. Secondary Outcome: Change From Baseline in Serum Immunoglobulin (Ig)G Concentration Over Time
Description: Change from baseline in serum immunoglobulin (Ig)G concentration over time was reported.
Time Frame: Baseline to Weeks 2, 4, 8, 12, 24, up to 253 days post-baseline, up to 257 days post-baseline
Population: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. Here, 'n' included the number of participants evaluated for specific timepoints. As per planned analysis, data is reported for individual arms and for all (total) participants both.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab | Nipocalimab (All Participants)
Number analyzed (Participants) | 5 | 27 | 32
g/L
  Week 2 | -6.888 (0.6104) | -5.457 (1.2510) | -5.681 (1.2804)
  Week 4: number analyzed (Participants) | 5 | 26 | 31
  Week 4 | -3.234 (1.1858) | -2.796 (0.9728) | -2.866 (1.0014)
  Week 8: number analyzed (Participants) | 5 | 19 | 24
  Week 8 | -2.996 (1.3773) | -3.122 (1.3466) | -3.095 (1.3235)
  Week 12: number analyzed (Participants) | 4 | 17 | 21
  Week 12 | -3.243 (1.6378) | -3.639 (2.2627) | -3.563 (2.1269)
  Week 24: number analyzed (Participants) | 1 | 5 | 6
  Week 24 | -3.870 (NA) — Here, NA indicates that standard deviation could not be calculated for 1 participant. | -4.072 (1.2826) | -4.038 (1.1502)
  253 days post-baseline: number analyzed (Participants) | 0 | 14 | 14
  253 days post-baseline |  | -3.494 (1.9208) | -3.494 (1.9208)
  257 days post-baseline: number analyzed (Participants) | 5 | 16 | 21
  257 days post-baseline | -1.150 (0.5687) | -0.020 (1.6162) | -0.289 (1.5056)

ADVERSE EVENTS:
Time Frame: Up to 257 days post-baseline (Day 1)
Description: The safety analysis set included all participants who received at least 1 dose of study drug nipocalimab.
Arm/Group | Placebo-Nipocalimab | Nipocalimab-Nipocalimab
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/30
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/30
Other Adverse Events (participants affected / at risk) | 4/7 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Nipocalimab (N=7) | Nipocalimab-Nipocalimab (N=30)
Coronavirus Infection (Infections and infestations) | 0 | 1
Covid-19 Pneumonia (Infections and infestations) | 1 | 0
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myasthenia Gravis (Nervous system disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Nipocalimab (N=7) | Nipocalimab-Nipocalimab (N=30)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 1
Conjunctival Hyperaemia (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Feeling Hot (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 3
Peripheral Swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1
Blood Immunoglobulin G Decreased (Investigations) | 1 | 4
Blood Potassium Decreased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 2
Neutrophil Count Increased (Investigations) | 0 | 2
Platelet Count Decreased (Investigations) | 0 | 1
White Blood Cell Count Increased (Investigations) | 0 | 1
Vitamin B6 Deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Myasthenia Gravis (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Depressed Mood (Psychiatric disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased Viscosity of Upper Respiratory Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was originally halted due to the COVID-19 pandemic. The study was later terminated prematurely due to the continuing COVID-19 pandemic, and because the participants will have the option to enter into an open-label extension portion of a planned future study. It was not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03896295/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03896295/SAP_001.pdf